CLINICAL TRIAL: NCT04336280
Title: The Prevalence and Clinical Presentation of Detrusor Underactivity and Its Urodynamic Characteristics
Brief Title: Detrusor Underactivity: Presentation and Urodynamic Characteristics
Status: Completed | Type: Observational
Sponsor: Mutah University (Other)
Collaborators: Istishari Urology Center (Unknown)
Responsible Party: Principal Investigator, Fadi Sawaqed, Assistant Professor, Mutah University
Other Study IDs: IUC - Detrusor Underactiivity
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Detrusor Underactivity
MeSH Terms: conditions — Urinary Bladder, Underactive | interventions — Urodynamics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Symptom questionnaire — Arabic version of the International Prostate Symptom Score: Known and validated questionnaire to quantify and qualify the severity of symptoms of the lower urinary tract
Diagnostic Test: Urodynamics — Urodynamics: the standard diagnostic tool, it includes invasive recording of the pressure that is produced when the bladder muscle contracts via pressure sensors introduced in the urinary bladder through special types of urethral catheters.

SUMMARY:
Detrusor underactivity (DU) is a known disease of the muscles of the urinary bladder that defined as a weak contraction of the muscle resulting in a failure to achieve complete bladder emptying. Recently, DU as a cause of Lower Urinary Tract Symptoms in both men and women has been increasingly gaining attention. There is a major issue in differentiation of underactive bladder symptoms and other causes of lower urinary tract symptoms such as detrusor hyperactivity and impaired contractility (DHIC), hypersensitive bladder (HSB), detrusor overactivity (DO), bladder outlet obstruction (BOO) and Dysfunctional Voiding (DV). Urodynamics (UDS) is the standard diagnostic tool, it includes invasive recording of the pressure that is produced when the bladder muscle contracts via pressure sensors introduced in the urinary bladder through special types of urethral catheters. This study aims to determine the prevalence of DU along with its symptomatic and urodynamics (UDS) characteristics of DU in Jordanian population through a retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent UDS from July 2016 to August 2019

Exclusion Criteria:

* Patients with neurogenic bladder (NB) due to known underlying neurological disease, history of open pelvic surgery or major abdominal surgery, or using indwelling catheters or clean intermittent catheterization (CIC).

Ages: 18 Years to 87 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study has reviewed a retrospective chart for 334 patients underwent UDS at the Istishari Urology Center (IUC), Amman, Jordan from July 2016 to August 2019.
  The study has excluded 77 records of patients in the initial stage either due to missing data (4 cases) or exclusion criteria (73 cases), the final study population was considered to be 206 patients.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of detrusor underactivity in Jordan | 3 years
  The proportion of patients with lower urinary tract symptoms found to be affected by Detrusor underactivity
Symptomatic presentation of Detrusor underactivity | over one month period prior to clinical evaluation during the 3 years time period
  Arabic version of the International Prostate Symptom Score was used to assess the prevalence and severity of the symptoms that are associated with detrusor underactivity. The questionnaire includes 8 questions, the 1st 7 questions are about the urinary symptoms (Incomplete emptying, urinary frequency, intermittency, urgency, weak urine stream, straining and nocturia) and the 8th is about Quality of Life due to Urinary Symptoms. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). The answers to the 8th question (quality of life) range from "delighted" to "terrible" or 0 to 6.
Urodynamics parameters | Each test takes around 30-45 minutes, all urodymanics studies were performed during the study period
  Urodynamics is a series of tests conducted in an outpatient setting that evaluates the function of the urinary bladder, including physiological parameters of how completely the bladder, sphincter and urethra are storing and releasing urine. These parameters are recorded by pressure sensors that are inserted into the bladder via special urinary catheters to measure the pressure that is generated during storing and releasing urine. The assessment of urodynamic variables is based on bladder capacity, presence of involuntary bladder muscle contractions, bladder volume at 1st sensation of bladder filling, bladder volumes at normal and strong desire for urination, detrusor pressure at maximum flow of urine during voiding, volume voided, and the post-void residual urine volume. All urodynamic testing was performed based on the International Continence Society standards.

CONTACTS AND LOCATIONS:
Locations (1):
- Istishari Urology Center (IUC), Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and analyzed during the current study are available from the corresponding author on reasonable request.